CLINICAL TRIAL: NCT01704092
Title: Dexmedetomidine's Cardiac and Cognitive Influence on Patients Undergoing Off-pump Coronary Artery Bypass Graft Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xin Chen, MD, Principal Investigator, Undergraduate, Huazhong University of Science and Technology
Other Study IDs: 2012001
Record Dates: First submitted 2012-10-01; First posted 2012-10-11 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples are drawn from patients recruited into the study. We planned to draw blood samples from patients with their consent through the central line.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group High-dose: Dexmedetomidine loading dose 1μg/kg Dexmedetomidine maintenance dose 0.6μg/kg/h
  Interventions: Drug: Dexmedetomidine
- Group Low-dose: Dexmedetomidine loading dose 0.6μg/kg Dexmedetomidine maintenance dose 0.3μg/kg/h
  Interventions: Drug: Dexmedetomidine
- Group Control: Dexmedetomidine loading dose and Dexmedetomidine maintenance dose were placed with the same amount of 0.9% saline as placebo
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine

SUMMARY:
The investigators hypothesized that dexmedetomidine as an anesthetic adjunct can be used in the setting of off-pump coronary bypass procedure and can provide benefits to cardiac function and cognitive performance on the ground of the dexmedetomidine's characteristics.

DETAILED DESCRIPTION:
The emergence of off-pump coronary artery bypass grafting (OPCAB) procedure brings up new challenges to anesthesiologists and urges us to contemplate the choice of anesthetics. In face of these challenges Dexmedetomdine with multiple unique traits can readily fit into this situation.

Off-pump coronary artery bypass (OPCAB) procedure is an emerging procedure which might bring benefit to patients in comparison with conventional CABGs although final words about outcomes haven't been reached on the basis of recent literature. However, OPCAB technique definitely requires more involvement of anesthesiologists especially in cases where hemodynamic compromise is usually inevitable during anastomosis of Lcx or PDA and early extubation in the OR is expected1. Thus, the investigators are encountered with more intraoperative challenges caused by OPCAB than routine CABGs. Concerning about challenges the investigators might take on, the investigators shall not only pay more attention to surgeons' manipulation but also review anesthetics that the investigators have selected to find an optimal plan to minimize adverse effects on heart and other important organs. With this perspective, dexmedetomidine come into our sight with its peculiar traits of hemodynamic effects and assumed cardiac protective effects.

Dexmedetomidine as a more selective α2-adrenoreceptor agonist than clonidine has gradually gain popularity in anesthetic and ICU settings for its unique pharmacologic characteristics. Dexmedetomidine provides sufficient sedative effects with minimal respiratory effect and then reduces the consumption of other sedative and antinociceptive drugs.Given specific requirements of OPCAB surgery, dexmedetomidine's may be more suitable in varying aspects. Firstly, dexmedetomine can dramatically diminish the level of serum catecholamine (CA). As the investigators know, the diminished level of catecholamine indicates less stress response to surgical stimuli and lower incidence of cardiac events. Secondly, the relatively slower HR by dexmedetomidine can decrease oxygen consumption of myocardium and consequently improve the perfusion of endangered ischemic area. In addition, the decreased HR which is assumably analogous to effects of esmolol or other β-blockers can reduce the occurrence of tachycardia and minimize the motion of heart when "bypass" procedure is performed on the target vessels. Thirdly, it has been reported that dexmedetomidine can alleviate sufferings of renal function during major thoracic surgery .Thus, it is implied that dexmedetomidine might in the similar way ameliorate the damage to renal system caused by hours of stress response and havoc of SIRS ,and then improve clinical prognosis . In view of assumptions the investigators have proposed on the ground of dexmedetomidine's characteristics and specific requirements of OPCAB surgery, the investigators are expecting that dexmdetomidine can fit the situation where patients' limited capacity of coronary artery and sophisticated pathophysiological courses have to be taken into account.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) scores are between classⅡand Ⅲ
* undergo off-pump coronary artery bypass grafting (OPCAB)

Exclusion Criteria:

* left ventricular ejection fraction <40%
* left ventricular aneurysm
* acute myocardial infarction in latest two weeks
* atrial fibrillation
* associated vascular diseases
* severe systemic diseases involving the renal and hepatic systems
* respiratory disease( forced vital capacity less than 50% of predicted values ) preoperative left bundle branch block .

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are planned to undergo off-pump coronary bypass surgery
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
cardioprective results represented by serial determination of troponin I (cTnI) cardioprective results represented by serial determination of troponin I (cTnI) | up to 3 days after the surgery
  The parameter measured is dynamic so that it is needed to detect the level at different time points
Hemodynamic values | from baseline to the end of the surgery
  On the basis of our experience, the period from baseline to the end of the surgery is five hours on average and would depend on the complexity of the surgical procedure
Serum level of β-amyloid protein | up to 3 days after the surgery
  The study is going to reflect the degree of central nerve system damage by detecting the level of S100 protein in serum. The serum level of S100 is preferred rather than the CSF sample because the approach of CSF sample obtaining is invasive and costly.
Serum level of S100 protein | up to 3 days after the surgical procedure
  The study is going to reflect the degree of central nerve system damage by detecting the level of S100 protein in serum. The serum level of S100 is preferred rather than the CSF sample because the approach of CSF sample obtaining is invasive and costly.

SECONDARY OUTCOMES:
intraoperative and postoperative urine output (UO), extubation time (ET), length of stay in ICU(LOSICU ) and length of hospital stay (LOS) | participants will be followed for the duration of hospital stay, an expected average of4 weeks
  The intraoperative and postoperative urine output (UO), extubation time (ET), length of stay in ICU(LOSICU ) are measured in ICU while the length of hospital stay is recorded at the discharge of every patient.
Mini-mental state examination(MMSE) scoring | up to patients' discharge from hospital
  The study is planned to detect the cognitive performance with this commonly used cognitive evaluation scoring

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology ,Tongji Hospital, Tongji Medical College,Huazhong University of Science and Technology, Wuhan, Hubei, China